CLINICAL TRIAL: NCT05303727
Title: Clinical Research of Allogeneic Hematopoietic Stem Cell Transplantation for Treatment of Children With Stage 4/M Neuroblastoma: A Prospective, Single-arm, Phase II, Multi-center Trial
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation for 4/M Neuroblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-126
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-03

CONDITIONS: Neuroblastoma
Keywords: allogeneic stem cell transplantation
MeSH Terms: conditions — Neuroblastoma | interventions — Antilymphocyte Serum; fludarabine; fludarabine phosphate; Cyclophosphamide; Topotecan; Melphalan; Thiotepa; Busulfan; Cyclosporine; Tacrolimus; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Intervention Model Description: There are 3 groups according to different sources of donor: (1) Cord blood HSCT: Flu+Bu+CTX+Topotecan (without ATG); (2) Peripheral blood HSCT or haploid bone marrow combined with peripheral stem cell transplantation: Flu+Bu+Melphalan+Antithymocyte globulin (ATG)+ Thiotepa (TT) or (3) Flu+Bu+Melphalan+ATG (applicable to peripheral stem cells or haploid bone marrow combined with peripheral stem cell transplantation for which TT cannot be used).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conditioning regimen for different sources of donors (Experimental): There are 3 groups according to different sources of donor: (1) Cord blood HSCT: Flu+Bu+CTX+Topotecan (without ATG); (2) Peripheral blood HSCT or haploid bone marrow combined with peripheral stem cell transplantation: Flu+Bu+Melphalan+Antithymocyte globulin (ATG)+ Thiotepa (TT) or (3) Flu+Bu+Melphalan+ATG (applicable to peripheral stem cells or haploid bone marrow combined with peripheral stem cell transplantation for which TT cannot be used).
  Interventions: Drug: Anti Thymocyte Globulin; Drug: Fludarabine; Drug: Cyclophosphamide injection; Drug: Topotecan; Drug: Melphalan; Drug: Thiotepa; Drug: Busulfan; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Methotrexate

INTERVENTIONS:
Drug: Anti Thymocyte Globulin — 2.5 mg/kg/day；2 doses on day -3 and day -2 for matched sibling donor transplantation；3 doses on day -4，-3 and day -2 for unrelated donor transplantation；4 doses on day -5，-4，-3 and day -2 for haploidentical donor transplantation
  Other Names: ATG
Drug: Fludarabine — 30 mg/m2/day for 5 days
  Other Names: Fludara
Drug: Cyclophosphamide injection — 60 mg/kg/day for 2 days in cord blood stem cell transplantation
  Other Names: CTX
Drug: Topotecan — 2mg/m2/day for 3 days in cord blood stem cell transplantation
  Other Names: Topotecan Hydrochloride
Drug: Melphalan — 70mg/m2/day，for peripheral stem cell transplantation or haploidentical bone marrow combined with peripheral stem cell transplantation；2 doses on day -3 and day -2 when conditioning regimen containing thiotepa；3 doses on day -4，-3 and day -2 when conditioning regimen not containing thiotepa；
  Other Names: Alkeran
Drug: Thiotepa — 5 mg/kg/day for 2 days in peripheral stem cell transplantation or haploidentical bone marrow combined with peripheral stem cell transplantation
  Other Names: thiophosphoramide
Drug: Busulfan — 0.8mg/kg/dose；8 doses in cord blood stem cell transplantation；12 doses in peripheral stem cell transplantation or haploidentical bone marrow combined with peripheral stem cell transplantation when conditioning regimen containing thiotepa；16 doses in peripheral stem cell transplantation or haploidentical bone marrow combined with peripheral stem cell transplantation when conditioning regimen not containing thiotepa；
  Other Names: Busulfex
Drug: Cyclosporine — 2.5~4 mg/kg/dose every 12 hours orally；1.5~2 mg /kg/dose every 12 hours intravenously; trough concentration maintained at 150~250ng/ml
  Other Names: Sandimmune
Drug: Tacrolimus — 0.02~0.03 mg/kg/day as continuous infusion or 12 hour divided doses
  Other Names: Prograf
Drug: Mycophenolate Mofetil — 15 mg/kg/dose every 12 hours
  Other Names: Cellcept
Drug: Methotrexate — 15 mg/m2/dose on d+1 and 10 mg/m2/dose on d+3，d+6 in peripheral stem cell transplantation
  Other Names: amethopterin

SUMMARY:
Neuroblastoma (NB) is the most common extracranial solid tumor of embryonal origin in children. According to the International Neuroblastoma Risk Group (INRG) staging criteria and the International Neuroblastoma Staging System (INSS) ，NB preoperative staging is divided into L1, L2, M and Ms stages, the postoperative staging is divided into 1 to 4 stages and 4s stage. Among them, 4/M stage is of the highest degree of malignancy and the worst prognosis. Despite the aggressive combination therapy, the 5-year survival rate (OS) is still less than 15%, and the 2-year relapse rate is 80%. Currently, no effective treatment is accessible for refractory/relapsed stage 4/M NB after completing conventional therapy.

In hematopoietic stem cell transplantation (HSCT) , conditioning regimen with high-dose radiotherapy and chemotherapy is implemented to eradicate tumor cells and abnormal clonal cells in the patient, block the pathogenesis, and restore the patient's hematopoietic and immune systems by transplanting normal hematopoietic stem cells. According to the source of hematopoietic stem cells, HSCT can be divided into two types: autologous hematopoietic stem cell transplantation (auto-HSCT) and allogeneic hematopoietic stem cell transplantation (allo-HSCT). It has been confirmed that benefiting from the graft versus tumor(GVT) effect, allo-HSCT can clear residual lesions in refractory/relapsed NB patients post-auto-HSCT，and prolong the survival time of patients. Our center has explored the conditioning regimen, treatment of residual tumor lesions before transplantation, and strategies to reduce transplantation-related death (TRM) and enhance the GVT effect. However, the sample size is small, and multicenter and larger sample size research are needed. This study will further observe the clinical efficacy and safety of allo-HSCT in the treatment of 4/M stage NB, and provide a new treatment method and option for 4/M stage NB.

DETAILED DESCRIPTION:
Purposes: To evaluate the efficacy and safety of allo-HSCT in children with stage 4/M high-risk NB through a multi-center prospective single-arm clinical research grouped according to different types of donors, graft sources, and stratified conditioning regimen.

Primary objectives: To evaluate the efficacy (3-year OS, EFS) of allo-HSCT in the treatment of children with stage 4/M NB through a multicenter prospective single-arm clinical study.

Secondary objectives:

1. To evaluate the safety of allo-HSCT in the treatment of children with stage 4/M NB [toxicity of conditioning regimen, engraftment rate, early transplantation-related mortality (<100d TRM), transplantation-related complications (VOD, thrombotic microangiopathy(TMA), acute/chronic graft-versus-host disease (GVHD), Epstein-Barr virus(EBV)/cytomegalovirus(CMV) viremia and EBV/CMV related diseases or other pathogenic infections, etc.];
2. Improvement and optimization of allo-HSCT conditioning regimen. Outline: This is a multicenter study. Conditioning regimen: There are 3 protocols according to different sources of donor: (1) Cord blood HSCT: Flu+Bu+cyclophosphamide (CTX)+Topotecan (without ATG); (2) Peripheral blood HSCT or haploid bone marrow combined with peripheral stem cell transplantation: Flu+Bu+Melphalan+Antithymocyte globulin (ATG)+ Thiotepa (TT) or (3) Flu+Bu+Melphalan+ATG (applicable to peripheral stem cells or haploid bone marrow combined with peripheral stem cell transplantation for which TT cannot be used).

Transplantation: Patients undergo cord blood stem cell or bone marrow or granulocyte colony stimulating factor (G-CSF) mobilized peripheral blood stem cell transplantation on day 0.

GVHD prophylaxis: Cyclosporine or tacrolimus combined with methotrexate is used for related matched transplantation, cyclosporine combined with mycophenolate mofetil for umbilical cord blood transplantation, and cyclosporine combined with mycophenolate mofetil and methotrexate for haploidentical transplantation to prevent GVHD.

After completion of transplantation, patients are followed periodically at least 3 years.

ELIGIBILITY:
1. Evaluation criteria for disease before and after transplantation:

1. Complete response (CR): all primary and metastatic lesions disappear, and neuron specific enolase (NSE), catecholamines and metabolites return to normal.
2. Very good partial response (VGPR): the primary tumor volume is reduced by 90% to 99%, all measurable metastases disappear, and NSE, catecholamines and metabolites return to normal; radionuclide bone scanned lesions can be positive (because bone metastases have not healed), but if an metaiodobenzylguanidine (MIBG) scan is performed, all lesions are negative.
3. Partial response (PR): The volume of all primary tumors and measurable metastases is reduced by more than 50%, the number of bone-positive lesions is reduced by more than 50%, and there is no more than one bone-positive site.
4. Mixed response (MR): no new lesions, the volume of any one or more measurable lesions decreases more than 50%, and the volume of any other one or more lesions decreases less than 50%, and volume of any existing lesions increases less than 25%.
5. No response (NR): There are no new lesions, and the volume of any existing lesions decreases less than 50% or increases less than 25%.
6. Progressive disease (PD): new lesions appear, the volume of existing measurable lesions increases more than 25%, and the bone marrow changes from negative to positive.

2. Inclusion Criteria: one of the following criteria (2), (3) or (4) must be met and all other criterions must be met at the same time:

1. Age≤18 years old;
2. After at least 7 courses of induction chemotherapy (surgical resection of the primary tumor or metastatic disease has been completed during the period), evaluation of disease is CR, tumor markers (blood NSE and urine VMA) and minimal residual disease by flow cytometry of bone marrow and peripheral blood are negative; the primary tumor has completed radiotherapy before HSCT;
3. For patients with PR or VGPR, tumor markers (blood NSE and urine VMA) and minimal residual disease by flow cytometry of bone marrow and peripheral blood are negative; the primary tumor and metastatic lesions have completed radiotherapy before HSCT;
4. Relapsed patients achieve CR/VGPR/PR after re-induction or salvage chemotherapy, tumor markers (blood NSE and urine VMA) and minimal residual disease by flow cytometry of bone marrow and peripheral blood are negative; the primary tumor and metastatic lesions have completed radiotherapy before HSCT;
5. Whole brain and whole spinal cord radiotherapy have completed before HSCT in patients with central invasion at onset;
6. The blood routine has generally returned to normal and there is no dysfunction of major organs such as the heart, liver, lung, and kidney;
7. The guardian/patient accept the treatment of this research, sign the informed consent, and complete the follow-up.

3. Exclusion Criteria: meeting one of the following criterions:

1. With severe cardiac insufficiency, cardiac ejection fraction (EF) is less than 50%; or severe cardiac disease, the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
2. With severe pulmonary insufficiency (severe obstructive and/or restrictive ventilation disorders), the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
3. With severe liver function impairment, ALT>5 times upper limit of normal, or total bilirubin>3 times upper limit of normal; the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
4. With severe renal insufficiency, creatinine>2 times upper limit of normal; or corrected creatinine clearance rate Ccr<50ml/min; the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
5. With severe active bleeding or severe active infection; the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
6. Allergic reactions or serious adverse reactions occurred in the previous use of conditioning regimen-related drugs, the patient can not tolerate the conditioning regimen according to the investigators' evaluation;
7. The guardian/patient cannot understand or comply with the treatment plan;
8. Other reasons for not being selected due to the investigator's evaluation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
overall survival(OS) at 3 year | 3 years post-HSCT
  From the date of day 0 of transplantation until the date of death from any cause
event free survival(EFS) at 3 year | 3 years post-HSCT
  Survival time from day 0 of transplantation to the occurrence of the first adverse event. Disease or treatment-related adverse events, such as tumor recurrence, implant failure, and death, are counted in this study; accidental deaths that assessed unrelated to the above factors are not included

SECONDARY OUTCOMES:
incidence of conditioning toxicity | 100 days post-HSCT
  Conditioning toxicity is graded according to the Common Terminology Criteria for Adverse Events(CTCAE Version 5.0)
incidence of donor engraftment | 100 days post-HSCT
  Donor engraftment represents donor cells replace at least 95% of recipient hematopoietic stem cells.
early transplant-related mortality | 100 days post-HSCT
  Death due to transplantation, excluding other causes such as disease progression or relapse.
incidence of sinusoidal obstruction syndrome | 3 years post-HSCT
  Sinusoidal obstruction syndrome is diagnosed according to classification from the European society for blood and marrow transplantation.
incidence of transplant associated thrombotic microangiopathy(TA-TMA) | 3 years post-HSCT
  TA-TMA is diagnosed according to the Jodele standard.
incidence of acute graft versus host disease | 100 days post-HSCT
  Acute graft versus host disease is diagnosed according to the modified Glucksberg grading standard.
incidence of infection | 3 years post-HSCT
  e.g. EBV/CMV viremia or related disease, bacteria/fungi /tuberculosis infection
incidence of chronic graft versus host disease | 3 years post-HSCT
  Chronic graft versus host disease is diagnosed according to the grading and scoring system recommended by the "Chinese Consensus on the Diagnosis and management of Chronic Graft-versus-Host Disease(2021)".

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Jianpei Fang, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pastor ER, Mousa SA. Current management of neuroblastoma and future direction. Crit Rev Oncol Hematol. 2019 Jun;138:38-43. doi: 10.1016/j.critrevonc.2019.03.013. Epub 2019 Apr 1. PMID 31092383
- [Background] Basta NO, Halliday GC, Makin G, Birch J, Feltbower R, Bown N, Elliott M, Moreno L, Barone G, Pearson AD, James PW, Tweddle DA, McNally RJ. Factors associated with recurrence and survival length following relapse in patients with neuroblastoma. Br J Cancer. 2016 Oct 25;115(9):1048-1057. doi: 10.1038/bjc.2016.302. Epub 2016 Oct 4. PMID 27701387
- [Background] Monclair T, Brodeur GM, Ambros PF, Brisse HJ, Cecchetto G, Holmes K, Kaneko M, London WB, Matthay KK, Nuchtern JG, von Schweinitz D, Simon T, Cohn SL, Pearson AD; INRG Task Force. The International Neuroblastoma Risk Group (INRG) staging system: an INRG Task Force report. J Clin Oncol. 2009 Jan 10;27(2):298-303. doi: 10.1200/JCO.2008.16.6876. Epub 2008 Dec 1. PMID 19047290
- [Background] Brodeur GM, Pritchard J, Berthold F, Carlsen NL, Castel V, Castelberry RP, De Bernardi B, Evans AE, Favrot M, Hedborg F, et al. Revisions of the international criteria for neuroblastoma diagnosis, staging, and response to treatment. J Clin Oncol. 1993 Aug;11(8):1466-77. doi: 10.1200/JCO.1993.11.8.1466. PMID 8336186
- [Background] Smith V, Foster J. High-Risk Neuroblastoma Treatment Review. Children (Basel). 2018 Aug 28;5(9):114. doi: 10.3390/children5090114. PMID 30154341
- [Background] London WB, Bagatell R, Weigel BJ, Fox E, Guo D, Van Ryn C, Naranjo A, Park JR. Historical time to disease progression and progression-free survival in patients with recurrent/refractory neuroblastoma treated in the modern era on Children's Oncology Group early-phase trials. Cancer. 2017 Dec 15;123(24):4914-4923. doi: 10.1002/cncr.30934. Epub 2017 Sep 8. PMID 28885700
- [Background] Matthay KK, Reynolds CP, Seeger RC, Shimada H, Adkins ES, Haas-Kogan D, Gerbing RB, London WB, Villablanca JG. Long-term results for children with high-risk neuroblastoma treated on a randomized trial of myeloablative therapy followed by 13-cis-retinoic acid: a children's oncology group study. J Clin Oncol. 2009 Mar 1;27(7):1007-13. doi: 10.1200/JCO.2007.13.8925. Epub 2009 Jan 26. PMID 19171716
- [Background] Ladenstein R, Potschger U, Pearson ADJ, Brock P, Luksch R, Castel V, Yaniv I, Papadakis V, Laureys G, Malis J, Balwierz W, Ruud E, Kogner P, Schroeder H, de Lacerda AF, Beck-Popovic M, Bician P, Garami M, Trahair T, Canete A, Ambros PF, Holmes K, Gaze M, Schreier G, Garaventa A, Vassal G, Michon J, Valteau-Couanet D; SIOP Europe Neuroblastoma Group (SIOPEN). Busulfan and melphalan versus carboplatin, etoposide, and melphalan as high-dose chemotherapy for high-risk neuroblastoma (HR-NBL1/SIOPEN): an international, randomised, multi-arm, open-label, phase 3 trial. Lancet Oncol. 2017 Apr;18(4):500-514. doi: 10.1016/S1470-2045(17)30070-0. Epub 2017 Mar 2. PMID 28259608
- [Background] Du H, Chen J, Qin M, Fang J, Li Z, Zhu Y, Sun X, Huang D, Yu J, Tang Y, Hu S, Li J, Zhang Z, Luan Z. Pediatric hematopoietic stem cell transplantation in China: Data and trends during 1998-2012. Pediatr Transplant. 2015 Aug;19(5):563-70. doi: 10.1111/petr.12525. Epub 2015 Jun 8. PMID 26058853
- [Background] Uemura S, Ishida T, Thwin KKM, Yamamoto N, Tamura A, Kishimoto K, Hasegawa D, Kosaka Y, Nino N, Lin KS, Takafuji S, Mori T, Iijima K, Nishimura N. Dynamics of Minimal Residual Disease in Neuroblastoma Patients. Front Oncol. 2019 Jun 4;9:455. doi: 10.3389/fonc.2019.00455. eCollection 2019. PMID 31214500
- [Background] Hirayama M, Azuma E, Araki M, Komada Y, Nakagawa A. Evidence of graft-versus-tumor effect in refractory metastatic neuroblastoma. Transplantation. 2006 Jul 15;82(1):142-4. doi: 10.1097/01.tp.0000225780.90991.49. No abstract available. PMID 16861958
- [Background] Marabelle A, Paillard C, Tchirkov A, Halle P, Chassagne J, Demeocq F, Kanold J. Graft-versus-tumour effect in refractory metastatic neuroblastoma. Bone Marrow Transplant. 2007 Jun;39(12):809-10. doi: 10.1038/sj.bmt.1705681. Epub 2007 Apr 23. No abstract available. PMID 17450181
- [Background] Matthay KK, Seeger RC, Reynolds CP, Stram DO, O'Leary MC, Harris RE, Selch M, Atkinson JB, Haase GM, Ramsay NK. Allogeneic versus autologous purged bone marrow transplantation for neuroblastoma: a report from the Childrens Cancer Group. J Clin Oncol. 1994 Nov;12(11):2382-9. doi: 10.1200/JCO.1994.12.11.2382. PMID 7964954
- [Background] Ladenstein R, Lasset C, Hartmann O, Klingebiel T, Bouffet E, Gadner H, Paolucci P, Burdach S, Chauvin F, Pinkerton R, et al. Comparison of auto versus allografting as consolidation of primary treatments in advanced neuroblastoma over one year of age at diagnosis: report from the European Group for Bone Marrow Transplantation. Bone Marrow Transplant. 1994 Jul;14(1):37-46. PMID 7951119
- [Background] Yi ES, Son MH, Hyun JK, Cho HW, Ju HY, Lee JW, Yoo KH, Sung KW, Koo HH. Predictors of survival in patients with high-risk neuroblastoma who failed tandem high-dose chemotherapy and autologous stem cell transplantation. Pediatr Blood Cancer. 2020 Feb;67(2):e28066. doi: 10.1002/pbc.28066. Epub 2019 Nov 17. PMID 31736249
- [Background] Haghiri S, Fayech C, Mansouri I, Dufour C, Pasqualini C, Bolle S, Rivollet S, Dumas A, Boumaraf A, Belhout A, Journy N, Souchard V, Vu-Bezin G, Veres C, Haddy N, De Vathaire F, Valteau-Couanet D, Fresneau B. Long-term follow-up of high-risk neuroblastoma survivors treated with high-dose chemotherapy and stem cell transplantation rescue. Bone Marrow Transplant. 2021 Aug;56(8):1984-1997. doi: 10.1038/s41409-021-01258-1. Epub 2021 Apr 6. PMID 33824435
- [Background] Park JR, Kreissman SG, London WB, Naranjo A, Cohn SL, Hogarty MD, Tenney SC, Haas-Kogan D, Shaw PJ, Kraveka JM, Roberts SS, Geiger JD, Doski JJ, Voss SD, Maris JM, Grupp SA, Diller L. Effect of Tandem Autologous Stem Cell Transplant vs Single Transplant on Event-Free Survival in Patients With High-Risk Neuroblastoma: A Randomized Clinical Trial. JAMA. 2019 Aug 27;322(8):746-755. doi: 10.1001/jama.2019.11642. PMID 31454045
- [Background] Milano F, Gooley T, Wood B, Woolfrey A, Flowers ME, Doney K, Witherspoon R, Mielcarek M, Deeg JH, Sorror M, Dahlberg A, Sandmaier BM, Salit R, Petersdorf E, Appelbaum FR, Delaney C. Cord-Blood Transplantation in Patients with Minimal Residual Disease. N Engl J Med. 2016 Sep 8;375(10):944-53. doi: 10.1056/NEJMoa1602074. PMID 27602666
- [Background] Chen YH, Xu LP, Liu DH, Chen H, Zhang XH, Han W, Wang FR, Wang JZ, Wang Y, Huang XJ, Liu KY. Comparative outcomes between cord blood transplantation and bone marrow or peripheral blood stem cell transplantation from unrelated donors in patients with hematologic malignancies: a single-institute analysis. Chin Med J (Engl). 2013 Jul;126(13):2499-503. PMID 23823825
- [Background] Eapen M, Rubinstein P, Zhang MJ, Stevens C, Kurtzberg J, Scaradavou A, Loberiza FR, Champlin RE, Klein JP, Horowitz MM, Wagner JE. Outcomes of transplantation of unrelated donor umbilical cord blood and bone marrow in children with acute leukaemia: a comparison study. Lancet. 2007 Jun 9;369(9577):1947-54. doi: 10.1016/S0140-6736(07)60915-5. PMID 17560447
- [Background] Rowinsky EK, Grochow LB, Hendricks CB, Ettinger DS, Forastiere AA, Hurowitz LA, McGuire WP, Sartorius SE, Lubejko BG, Kaufmann SH, et al. Phase I and pharmacologic study of topotecan: a novel topoisomerase I inhibitor. J Clin Oncol. 1992 Apr;10(4):647-56. doi: 10.1200/JCO.1992.10.4.647. PMID 1312588
- [Background] Cohn SL, Pearson AD, London WB, Monclair T, Ambros PF, Brodeur GM, Faldum A, Hero B, Iehara T, Machin D, Mosseri V, Simon T, Garaventa A, Castel V, Matthay KK; INRG Task Force. The International Neuroblastoma Risk Group (INRG) classification system: an INRG Task Force report. J Clin Oncol. 2009 Jan 10;27(2):289-97. doi: 10.1200/JCO.2008.16.6785. Epub 2008 Dec 1. PMID 19047291
- [Background] Sottile F, Gnemmi I, Cantilena S, D'Acunto WC, Sala A. A chemical screen identifies the chemotherapeutic drug topotecan as a specific inhibitor of the B-MYB/MYCN axis in neuroblastoma. Oncotarget. 2012 May;3(5):535-45. doi: 10.18632/oncotarget.498. PMID 22619121
- [Background] Rujkijyanont P, Photia A, Traivaree C, Monsereenusorn C, Anurathapan U, Seksarn P, Sosothikul D, Techavichit P, Sanpakit K, Phuakpet K, Wiangnon S, Chotsampancharoen T, Chainansamit SO, Kanjanapongkul S, Meekaewkunchorn A, Hongeng S. Clinical outcomes and prognostic factors to predict treatment response in high risk neuroblastoma patients receiving topotecan and cyclophosphamide containing induction regimen: a prospective multicenter study. BMC Cancer. 2019 Oct 16;19(1):961. doi: 10.1186/s12885-019-6186-z. PMID 31619207
- [Background] London WB, Frantz CN, Campbell LA, Seeger RC, Brumback BA, Cohn SL, Matthay KK, Castleberry RP, Diller L. Phase II randomized comparison of topotecan plus cyclophosphamide versus topotecan alone in children with recurrent or refractory neuroblastoma: a Children's Oncology Group study. J Clin Oncol. 2010 Aug 20;28(24):3808-15. doi: 10.1200/JCO.2009.27.5016. Epub 2010 Jul 26. PMID 20660830
- [Background] Kasow KA, Stewart CF, Barfield RC, Wright NL, Li C, Srivastava DK, Leung W, Horwitz EM, Bowman LC, Handgretinger R, Hale GA. A phase I/II study of CY and topotecan in patients with high-risk malignancies undergoing autologous hematopoietic cell transplantation: the St Jude long-term follow-up. Bone Marrow Transplant. 2012 Nov;47(11):1448-54. doi: 10.1038/bmt.2012.51. Epub 2012 Mar 19. PMID 22426752
- [Background] Philip T, Ladenstein R, Lasset C, Hartmann O, Zucker JM, Pinkerton R, Pearson AD, Klingebiel T, Garaventa A, Kremens B, Bernard JL, Rosti G, Chauvin F. 1070 myeloablative megatherapy procedures followed by stem cell rescue for neuroblastoma: 17 years of European experience and conclusions. European Group for Blood and Marrow Transplant Registry Solid Tumour Working Party. Eur J Cancer. 1997 Oct;33(12):2130-5. doi: 10.1016/s0959-8049(97)00324-9. PMID 9516868
- [Background] Kreissman SG, Seeger RC, Matthay KK, London WB, Sposto R, Grupp SA, Haas-Kogan DA, Laquaglia MP, Yu AL, Diller L, Buxton A, Park JR, Cohn SL, Maris JM, Reynolds CP, Villablanca JG. Purged versus non-purged peripheral blood stem-cell transplantation for high-risk neuroblastoma (COG A3973): a randomised phase 3 trial. Lancet Oncol. 2013 Sep;14(10):999-1008. doi: 10.1016/S1470-2045(13)70309-7. Epub 2013 Jul 25. PMID 23890779